CLINICAL TRIAL: NCT02512120
Title: Comparison of Volume Controlled Ventilation(VCV) vs Autoflow-volume Controlled Ventilation(Autoflow-VCV) During Robot-assisted Laparoscopic Radical Prostatectomy
Brief Title: Volume Controlled Ventilation vs Autoflow-volume Controlled Ventilation
Acronym: VCVAFVCV
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The backgroud of this study was not well discussed.
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Hye-Won Shin, Director, MD, PhD, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Autoflow46
Record Dates: First submitted 2015-07-29; First posted 2015-07-30 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- volume controlled ventilation (Experimental): Randomized 23 patients will be applied VCV during RALP.
  Interventions: Device: volume controlled ventilation
- autoflow-volume controlled ventilation (Active Comparator): Randomized 23 patients will be applied autoflow-VCV during RALP.
  Interventions: Device: autoflow-volume controlled ventilation

INTERVENTIONS:
Device: volume controlled ventilation — After induction of anesthesia and intubation, patients will be applied VCV by Zeus®(Dräger, Germany).
  - Tidal volume : 8ml/kg(ieal body weight), inspiration:expiration ratio = 1:2, FiO2 = 0.5, fresh gas flow = 3L/min respiratory rate(RR) : 12/min. After position, RR can changed 2 times each per 5 minutes to maintain end tidal CO2 around 35. Positive end expiratory pressure will not used.
  Arms: volume controlled ventilation
Device: autoflow-volume controlled ventilation — After induction of anesthesia and intubation, patients will be applied autoflow- VCV by Zeus®(Dräger, Germany).
  - Tidal volume : 8ml/kg(ideal body weight), inspiration:expiration ratio = 1:2, FiO2 = 0.5, fresh gas flow = 3L/min respiratory rate(RR) : 12/min. After position, RR can changed 2 times each per 5 minutes to maintain end tidal CO2 around 35. Positive end expiratory pressure will not used.
  Arms: autoflow-volume controlled ventilation

SUMMARY:
Volume controlled ventilation(VCV) is a most common used ventilation mode during general anesthesia. But VCV can cause high airway peak pressure when patient under steep Trendelenberg position with pneumoperitoneum. Autoflow-VCV can reduce airway peak pressure and improve dynamic compliance. We will compare parameters(arterial blood gas analysis, airway compliance, etc) when each group applied VCV and autoflow-VCV during RALP.

DETAILED DESCRIPTION:
Robot assisted laparoscopic radical prostatectomy(RALP) has been used to treatment of prostate cancer since 2001. RALP offers some advantage such as reduced blood loss, sparing nerves, less postoperative pain. However, RALP require steep Trendelenberg position with pneumoperitoneum. It can cause increased airway peak pressure and unwanted hemodynamic effect under conventional volume controlled ventilation(VCV). Autoflow-VCV use decelerating flow, can reduce airway peak pressure and improve dynamic compliance.

We will compare parameters(arterial blood gas analysis, airway compliance, etc) when each group applied VCV and autoflow-VCV during RALP.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age 19-65)
* American Society of Anesthesiology Classification I-III

Exclusion Criteria:

* cardiovascular disease, cerebrovascular disease, pulmonary disease
* over BMI 30

Ages: 19 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-08; Primary Completion 2016-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Airway pressure | 4hours
  Airway pressure will be measured under specified ventilation mode.

SECONDARY OUTCOMES:
Vital sign | 4hours
  Vital sign will be measured under specified ventilation mode.

OTHER OUTCOMES:
Arterial blood gas analysis | 4hours
  Arterial blood gas analysis will be measured under specified ventilation mode.

CONTACTS AND LOCATIONS:
Overall Officials: Hye-Won Shin, MD, PhD, Study Director — Department of anesthesiology and pain medicine, Korea University Anam Hospital